## Statistical Analysis Plan

Activated Macrophages and Ozone Toxicity

NCT02673775

June 7, 2023

**Primary Outcome Measure:** Concentrations of M1 and M2 macrophages in the sputum 24 hours after exposure.

Measure Description: The relative concentrations of M1 and M2 macrophages in the induced sputum sample will be assessed.

Statistical method: A paired t-test, with ratio of M2 to M1 macrophages in the induced sputum sample as the dependent variable, was used to compare the effect of ozone and clean air 24 hours after exposure. The level of significance ( $\alpha$ ) was set to 0.05.

**Primary Outcome Measure:** Concentrations of M1 and M2 macrophages in the sputum 48 hours after exposure.

Measure Description: The relative concentrations of M1 and M2 macrophages in the induced sputum sample will be assessed.

Statistical method: A paired t-test, with ratio of M2 to M1 macrophages in the induced sputum sample as the dependent variable, was used to compare the effect of ozone and clean air 48 hours after exposure. The level of significance ( $\alpha$ ) was set to 0.05.

**Primary Outcome Measure:** Concentrations of M1 and M2 macrophages in the sputum 72 hours after exposure.

Measure Description: The relative concentrations of M1 and M2 macrophages in the induced sputum sample will be assessed.

Statistical method: A paired t-test, with ratio of M2 to M1 macrophages in the induced sputum sample as the dependent variable, was used to compare the effect of ozone and clean air 72 hours after exposure. The level of significance ( $\alpha$ ) was set to 0.05.